CLINICAL TRIAL: NCT01076946
Title: Insights in the Pathophysiology of Transient Left Ventricular Ballooning Syndrome (TLVBS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: UZ Leuven, Department Interventional Cardiology
Other Study IDs: pathophysiology TLVBS
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2009-12

CONDITIONS: Transient Left Ventricular Ballooning Syndrome
Keywords: ballooning; TLVBS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TLVBS: patients with transient left ventricular ballooning

SUMMARY:
Transient left ventricular ballooning syndrome (TLVBS) is a cardiac syndrome that is characterised by acute but transient left ventricular (LV) dysfunction.

Since the syndrome clearly is not a rare phenomenon and since prognosis is not as benign as originally thought, there is a need for further research into the etiology and pathophysiology of TLVBS. Therefore the investigators aim to study the microvascular and endothelial function in their population of TLVBS patients.

DETAILED DESCRIPTION:
It was shown recently that in patients with previous TLVBS a cold pressor test (CPT) was able to induce new mid-ventricular and apical wall motion abnormalities, similar to those in the acute phase of the syndrome. Moreover, coronary blood flow (CBF), assessed by means of myocardial contrast echocardiography (MCE), increased in a group of control subjects but not in the TLVBS patients, suggesting a chronic impairment of coronary vasodilation reserve and thus microvascular dysfunction.

Since the syndrome clearly is not a rare phenomenon and since prognosis is not as benign as originally thought, there is a need for further research into the etiology and pathophysiology of TLVBS. Therefore the investigators aim to study the microvascular and endothelial function in their population of TLVBS patients. The project will be split up into two parts:

1. From the patients that are already known in the prospective registry, patients willing to participate after informed consent will be asked to undergo a "reactive hyperaemia - pulse amplitude tonometry" (RH-PAT) baseline and after CPT and a cardiac magnetic resonance scan (CMR), at least 3 months after the last TLVBS event.

   The RH-PAT evaluates endothelial function. The CMR-evaluation at rest consists of assessment of global and regional left ventricular function, the exclusion of irreversible damage (lack of gadolinium hyperenhancement) and the evaluation of rest perfusion. Subsequently, adenosine-induced hyperemia is induced by an infusion of 140 µg/kg/min adenosine for 3 to 4 minutes, with stress perfusion sequence starting at 3 minutes. After approximately 10 minutes, a CPT will be performed (180 seconds immersion of the left foot in ice water (4°C)) immediately followed by a series of CMR cine sequences and a second stress perfusion CMR sequence. Afterwards the RH-PAT examination is repeated and blood sampling will be done for measuring plasma levels of B-type natriuretic peptide (BNP), the catecholamines epinephrine, norepinephrine, and dopamine and a marker for endothelial function endothelin-1.

   Patients will be monitored for one hour and before discharge two-dimensional (2D) echocardiography will be performed to exclude residual wall motion abnormalities. The investigators goal is to include at least 30 patients in this protocol.
2. Patients who are newly admitted with TLVBS will follow a clinical path during index hospitalisation including serial ECG recording, serial blood sampling of cardiac biomarkers (Troponin I, CKMB), a sole sampling of BNP, catecholamines and endothelin-1, a RH-PAT measurement, a 2D echocardiogram, a coronary angiogram and a CMR with rest perfusion sequence. They will also be asked to return to the hospital at 3 months for the evaluation mentioned above. Patients will be added to the prospective registry.

ELIGIBILITY:
Inclusion Criteria:

* For filling criteria of TLVBS
* Presence of acute or subacute cardiac symptoms or events - Presence of reversible balloon-like left ventricular (LV) wall motion abnormalities (WMAs) that extend beyond the vascular distribution of a single epicardial vessel
* Absence of ≥ 50% luminal narrowing or acute plaque rupture or intracoronary thrombus in the left anterior descending artery (LAD) in case the LAD extends well beyond the LV apex
* Absence of pheochromocytoma, myocarditis, recent cardiac events or procedures, and recent stroke or head injury
* Signed informed consent

Exclusion Criteria:

* Not complying with any or more of the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients that were or will be admitted with TLVBS
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kayaert, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium